CLINICAL TRIAL: NCT00652470
Title: International Infant Hydrocephalus Study: A Multicentre, Prospective Study
Brief Title: A Study Comparing Two Treatments for Infants With Hydrocephalus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: The International Study Group for Neuroendoscopy (ISGNE) (Unknown); The International Society for Pediatric Neurosurgery (Other)
Responsible Party: Principal Investigator, Abhaya Kulkarni, Staff neurosurgeon, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1000007601
Record Dates: First submitted 2008-03-31; First posted 2008-04-03 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Hydrocephalus
Keywords: infants; Hydrocephalus; Cerebrospinal Fluid Shunt; Ventriculostomy; neurosurgery
MeSH Terms: conditions — Hydrocephalus | interventions — Ventriculostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ETV (Active Comparator)
  Interventions: Procedure: Endoscopic Third Ventriculostomy
- CSF Shunt (Active Comparator)
  Interventions: Procedure: CSF Shunt Insertion

INTERVENTIONS:
Procedure: Endoscopic Third Ventriculostomy — A standard frontal burr hole will be made and an endoscopic camera used to visualize the floor of the third ventricle. A ventriculostomy will be created in the floor of the third using the surgeon's own preferred method of perforation.
  Arms: ETV
Procedure: CSF Shunt Insertion — The procedure involves creating a burr hole in the frontal or occipital regions and cannulating the ventricle with a silastic catheter. This is then attached to a valve mechanism and distal silastic tubing which runs subcutaneously in the peritoneal cavity.
  Arms: CSF Shunt

SUMMARY:
The purpose of this study is to study whether infants with triventricular hydrocephalus (TVH) have a better long-term outcome at 5 years when they are treated with a new procedure, endoscopic third ventriculostomy (ETV), than infants treated with the more traditional treatment, insertion of a cerebrospinal fluid (CSF) shunt.

DETAILED DESCRIPTION:
TVH is a relatively uncommon condition in infants, in which CSF accumulates in the brain's ventricles due to a blockage in outflow at the level of cerebral aqueduct. This can cause increased intracranial pressure, with adverse effect on brain development. The causes of this include congenital aqueductal stensois or acquired aqueductal stenosis from previous brain hemorrhage or infection.

TVH is currently treated through one of the following two approaches:

* Extra-cranial CSF diversion through ventricular shunts. Extra-cranial shunting has been the standard approach over the past few decades, since functional shunts were first developed and inserted successfully.
* Intra-cranial internal CSF diversion using endoscopic techniques. The principles of internal diversion were clear from the time neurosurgeons first understood the nature of hydrocephalus. However, internal diversion was never really practical or successful on a large scale until the more recent development of neuroendoscopy. There is currently a revived interest in diversionary hydrocephalus treatment through neuroendoscopic surgical techniques, with the primary focus on endoscopic third ventriculostomy (ETV).

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic TVH requiring treatment.
* No previous treatment for TVH
* Under 24 months of age at time of surgery
* Full-term pregnancy (>36 weeks)
* Mandatory pre-operative MRI that includes mid-sagittal T1 & T2 scans which show: Tri-ventricular pattern of hydrocephalus; proof of no flow through aqueduct; presence of CSF collection over the convexity and/or inter-hemispheric fissure is acceptable; configuration of third ventricle floor could vary; deformed tectal plate is acceptable; posterior fossa fluid collections may be included as long as: aqueduct is closed; vermis preserved (complete Dandy Walker Syndrome excluded); questionable flow in aqueduct acceptable as long as TVH exists
* History or suggestion of intra-ventricular bleed (intra-uterine or post-natal) or intracranial infection qualifies (excluding intraventricular hemorrhage of prematurity).
* Ability to participate in followup for at least 5 years

Exclusion Criteria:

* Open Spina Bifida
* Complete Dandy Walker syndrome (vermian agenesis / dysgenesis)
* Prematurity
* Perinatal asphyxia
* Severe dysmorphic anatomical features or known chromos (e.g. agenesis of corpus callosum, heterotopias, large cysts)
* intracranial tumor

Ages: 1 Day to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 182 (Estimated)
Dates: Start 2005-09; Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Health Status Outcome as measured by the Health Utilities Index - 2 | At 5 years of age

SECONDARY OUTCOMES:
Death | Duration of the Study
Neurodevelopment as measured by the Denver Developmental Screening Test | Up to 3 years of Age
Health status outcome using the Hydrocephalus Outcome Questionnaire | At 5 years of Age
In-depth Evaluation of Neurodevelopment, Functioning and Intelligence, as mesured by the Weschler Intelligence Scale for Children or Weschler Preschool and Primary Scale of Intelligence | At 5 years of Age
Number of Subsequent Hydrocephalus-Related Operations | Duration of the Study
Surgical Morbidity | Duration of the Study
Incidence of failure of initial intervention | Duration of the Study
Hospitalization Time | 5 years post-operation
Need for repeat radiological scans | Duration of the Study
Complications such as CNS infection, focal neurological deficit, significant hemorrhage, seizures requiring medication | Duration of the Study
Ventricular size and the existence of flow void (ETV group)assessed through radiological evaluation | 3 years of age

CONTACTS AND LOCATIONS:
Overall Officials: Abhaya Kulkarni, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada; Shlomi Constantini, MD, Principal Investigator — Dana Children's Hospital, Tel Aviv Medical Center; Spyros Sgouros, MD, Principal Investigator — Birmingham Children's Hospital
Locations (22):
- Children's Medical Center of Dallas, Dallas, Texas, United States
- Nacional de Pediatria, Buenos Aires, Argentina
- Brazil (2):
  - Biocor Instituto, Nova Lima
  - UNIFESP, São Paulo
- The Hospital for Sick Children, Toronto, Ontario, Canada
- University Hospital Gießen and Marburg, Giessen, Germany
- University of Debrecen, Debrecen, Hungary
- India (2):
  - Sanjay Gandhi Postgraduate Institute of Medical Sciences, Lucknow
  - All India Institute of Medical Sciences, New Delhi
- Dana Children's Hospital, Tel Aviv Medical Center, Tel Aviv, Israel
- Italy (2):
  - Giannina Gaslini Hospital, Genova
  - Catholic University Medical School Rome, Rome
- University Medical Center St Radboud, Nijmegen, Netherlands
- Poland (3):
  - Medical University of Silesia, Katowice
  - Polish Mother's Memorial Hospital, Lodz
  - Children's Memorial Health Institute, Warsaw
- Burdenko Neurosurgical Institute, Moscow, Russia
- Institute for Neurosurgery, Belgrade, Serbia
- Hospital Sant Joan de Deu, Barcelona, Spain
- Hacettepe University Hospital, Ankara, Turkey (Türkiye)
- United Kingdom (2):
  - Birmingham Children's Hospital, Birmingham
  - Alder Hey Children's Hospital, Liverpool

REFERENCES:
- [Derived] Kulkarni AV, Sgouros S, Leitner Y, Constantini S; International Infant Hydrocephalus Study Investigators. International Infant Hydrocephalus Study (IIHS): 5-year health outcome results of a prospective, multicenter comparison of endoscopic third ventriculostomy (ETV) and shunt for infant hydrocephalus. Childs Nerv Syst. 2018 Dec;34(12):2391-2397. doi: 10.1007/s00381-018-3896-5. Epub 2018 Jul 9. PMID 29987375
- [Derived] Kulkarni AV, Sgouros S, Constantini S; International Infant Hydrocephalus Study Investigators. Outcome of treatment after failed endoscopic third ventriculostomy (ETV) in infants with aqueductal stenosis: results from the International Infant Hydrocephalus Study (IIHS). Childs Nerv Syst. 2017 May;33(5):747-752. doi: 10.1007/s00381-017-3382-5. Epub 2017 Mar 29. PMID 28357554
- [Derived] Kulkarni AV, Sgouros S, Constantini S; IIHS Investigators. International Infant Hydrocephalus Study: initial results of a prospective, multicenter comparison of endoscopic third ventriculostomy (ETV) and shunt for infant hydrocephalus. Childs Nerv Syst. 2016 Jun;32(6):1039-48. doi: 10.1007/s00381-016-3095-1. Epub 2016 Apr 23. PMID 27107887